CLINICAL TRIAL: NCT02404623
Title: The Effect of Vitamin D Administration to Premature Infants on Vitamin D Status and Respiratory Morbidity During the First Year of Life
Brief Title: The Effect of Vitamin D Administration to Premature Infants on Vitamin D Status and Respiratory Morbidity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Principal Investigator, Inbal Golan- Tripto MD, Pediatrics pulmonologist, Soroka University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SOR -0292-14-CTIL
Record Dates: First submitted 2015-03-18; First posted 2015-03-31 (Estimated); Last update posted 2018-02-14 (Actual); Status verified 2018-02

CONDITIONS: Other Preterm Infants; Vitamin D Deficiency; Bronchiolitis; Asthma; Pneumonia
Keywords: Vitamin D; Respiratory Morbidity; prematurity
MeSH Terms: conditions — Vitamin D Deficiency; Bronchiolitis; Asthma; Pneumonia; Premature Birth | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Group (Experimental): 800 IU of Vitamin D once daily
  Interventions: Dietary Supplement: Vitamin D
- Control Group (Other): 400 IU of Vitamin D once daily, the standard of care
  Interventions: Dietary Supplement: Vitamin D

INTERVENTIONS:
Dietary Supplement: Vitamin D — also known as Cholecalciferol, is one of the two most important compounds within the group of Vitamin D. It can be ingested from the diet and from supplements. In this study it is pharmacologically acquired and referred to as Vitamin D

SUMMARY:
This trial objective is to assess whether doubling the daily intake of vitamin D improves serum vitamin D levels and serves as primary prevention of respiratory infections and asthma in premature infants.

This is a prospective randomized (1:1) double-blinded trial.

The study population will be randomized into two groups (1:1):

* Intervention Group - 800 IU of Vitamin D once daily
* Control Group - 400 IU of Vitamin D once daily Patients will be followed up for one year after randomization for serum Vitamin D levels and respiratory morbidity.

DETAILED DESCRIPTION:
The rational of this trial is that a daily supplementation of a double dose of Vitamin D (800 IU instead of 400 IU) to late premature infants during the first year of life will result in elevated Vitamin D serum levels and in an improvement in respiratory morbidity.

This randomized trial of vitamin D supplementation is planned to determine the optimal dose of daily vitamin D supplementation required to achieve sufficient vitamin D levels in preterm infants and to assess whether doubling the daily intake of vitamin D may serve as primary prevention of respiratory infections and asthma in premature infants.

ELIGIBILITY:
Inclusion Criteria:

1. Preterm infant born at 32+6 to 36+6 weeks of gestational age
2. Born at Soroka University Medical Center
3. Signed informed consent
4. Participants in the trial will be insured by "Clalit" HMO

Exclusion Criteria:

1. Chromosomal abnormality
2. Neurological or muscular congenital anomalies
3. Congenital cardiac defect
4. Congenital respiratory anomalies
5. Congenital GIT/ liver/ renal anomalies that effect the absorption and/or metabolism of Vitamin D and/or other substances.
6. Admission after birth to NICU persists more than 5 days

Ages: 33 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2015-04; Primary Completion 2018-02-12 (Actual); Study Completion 2018-02-12 (Actual)

PRIMARY OUTCOMES:
Improved serum vitamin D levels in the intervention group (receiving 800 IU daily) in comparison to the control group (receiving 400 IU daily) | 12 months of age

SECONDARY OUTCOMES:
respiratory morbidity prevalence | first year
  Reports given by the parents via questionnaire at 3, 6, 9 and 12 months.
respiratory morbidity prevalence | first year
  Information collected from medical records containing the data of diagnosis or admission to pediatrics departments due to: bronchiolitis, wheezing, upper or lower respiratory tract infections, asthma and pneumonia
respiratory morbidity prevalence | first year
  Information collected from medical records containing the data of medication consumption such as bronchodilators, inhaled corticosteroid, systemic corticosteroids (along with respiratory disease) and antibiotics (along with respiratory infection).

CONTACTS AND LOCATIONS:
Overall Officials: Inbal Golan Tripto, MD, Principal Investigator — Soroka University Medical Center
Locations (1):
- Soroka University Medical Center, Beersheba, P.O.Box 151, Israel

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Huey SL, Acharya N, Silver A, Sheni R, Yu EA, Pena-Rosas JP, Mehta S. Effects of oral vitamin D supplementation on linear growth and other health outcomes among children under five years of age. Cochrane Database Syst Rev. 2020 Dec 8;12(12):CD012875. doi: 10.1002/14651858.CD012875.pub2. PMID 33305842